CLINICAL TRIAL: NCT00541216
Title: Ephedrine for the Treatment of Congenital Myasthenia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ephedrine-hmo-ctil
Record Dates: First submitted 2007-10-07; First posted 2007-10-10 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Myasthenic Syndromes, Congenital
Keywords: congenital myasthenia; ephedrine
MeSH Terms: conditions — Myasthenic Syndromes, Congenital | interventions — Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ephedrine

SUMMARY:
Previous research has demonstrated possible efficacy of Ephedrine in the treatment of congenital myasthenia caused by end-plate acetylcholinesterase deficiency.

The aim of the current study is to test the hypothesis that Ephedrine may be beneficial to these patients.

To test this hypothesis we will perform a double blind, placebo-controlled, crossover study clinical efficacy and safety study.

Drug naïve patients who agree to participate will be randomized to two groups. Each group will be treated in a blinded manner for 5 weeks with either placebo or Ephedrine HCl in an escalating dose up to 100 mg per day divided in two doses. After five weeks the groups will cross over and continue treatment or placebo for a further five weeks.

Evaluations of strength and fatiguability will be done at baseline, at the end of each five week period and after a further two weeks.

Safety will be assessed weekly by the investigators using interview and physical examination.

Outcome measures will include Barthel index, Quality of life questionnaire, Timed up and go, spirometry, timed elevation of limbs, and force measurements.

All patients will report to the clinic as per study schedule (See Appendix A). Specifically, the 12 clinic visits will include: baseline (1), safety and efficacy assessments(10) and closeout (1).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients , with congenital myasthenia, belonging to a previously reported kindred diagnosed with COLQ deficiency.

Exclusion Criteria:

* History of allergy to Ephedrine or any inactive component.
* Significant abnormalities in screening Cardiovascular parameters (blood pressure, pulse).
* Surgery within 6 weeks of screening.
* Concurrent use of any other medication except steroids.
* Pregnancy.
* Thyrotoxicosis.
* Co-morbid conditions or other neurological disorders that would confound assessment of clinical parameters.
* Participation in another clinical trial within 30 days of study start.
* Patients who are non-cooperative or parents/ legal guardians who are unwilling to sign consent form.

Ages: 12 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-10

PRIMARY OUTCOMES:
strength and fatiguability: walking, straight arm raising, spirometry. | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simon Edvardson, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel